CLINICAL TRIAL: NCT01991366
Title: Should Integrilin be an Integral Part of Adjunctive Therapy in Patients Undergoing Primary Percutaneous Coronary Intervention for ST-Elevation Myocardial Infarction?
Brief Title: Should Integrilin be an Integral Part of Adjunctive Therapy in Patients Undergoing Primary PCI for ST-Elevation MI?
Status: Withdrawn | Type: Observational
Why Stopped: lack of funding
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Integrilin Stemi
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: ST-elevation Myocardial Infarction; Acute Myocardial Infarction
Keywords: Major adverse microvascular integrity; all cause mortality; Q Wave MI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Eptifibatide Pre PCI: Receive eptifibatide pre PCI
- Eptifibatide during PCI: Receive eptifibatide during PCI
- No Eptifibatide: Receive no eptifibatide

SUMMARY:
The aim of this observational study is to evaluate the in hospital and 6 month outcomes of the use of Glycoprotein IIb/IIIa inhibitor eptifibatide as adjunctive therapy in patients undergoing primary Percutaneous Coronary Intervention for ST-elevation myocardial infarction in a large tertiary referral center.

It is hypothesized that Glycoprotein IIb/IIIa inhibitor use during primary Percutaneous Coronary Intervention for ST-elevation myocardial infarction/ acute myocardial infarction is superior to unfractionated heparin alone or bivalirudin alone. Additionally, after propensity matching this superiority remains.

DETAILED DESCRIPTION:
This is a retrospective, observational, data analysis of approximately 800 patients who underwent primary Percutaneous Coronary Intervention at our institution since September 2000. Patients will have either received eptifibatide pre-or during Percutaneous Coronary Intervention or have received no eptifibatide. Patients who received a thrombolytic prior to Percutaneous Coronary Intervention will be excluded.

This analysis is estimated to take 1-2 months.

ELIGIBILITY:
Inclusion Criteria:

* Underwent Percutaneous Coronary Intervention at Washington Hospital Center since September 2000
* Either received eptifibatide pre-or during PCI or have received no eptifibatide.

Exclusion Criteria:

* Patients who received a thrombolytic prior to Percutaneous Coronary Intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent primary Percutaneous Coronary Intervention at Washington Hospital Center since September 2000 and received eptifibatide pre-or during PCI or have received no eptifibatide.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-10 (Estimated); Primary Completion 2014-10 (Estimated); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
All-cause mortality and composite or Q-wave myocardial infarction | Chart review 6 months after PCI
  6-month rates of all-cause mortality and the composite of all-cause mortality or Q-wave myocardial infarction.

SECONDARY OUTCOMES:
TIMI major bleeding | During hospital stay; average stay is less than 48 hours
  Thrombolysis In Myocardial Infarction (TIMI) major bleeding during hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States